CLINICAL TRIAL: NCT02274545
Title: Phase 1 Evaluation of the Safety and Immunogenicity of Live Influenza A Vaccine H7N9 (6-2) AA ca Recombinant (A/Anhui/1/2013 (H7N9) x A/Ann Arbor/6/60 ca), a Live Attenuated Virus Vaccine Candidate for Prevention of Influenza H7N9 Disease in 50 to 70 Year Olds in the Event of a Pandemic
Brief Title: Evaluating the Safety and Immunogenicity of a H7N9 Vaccine for the Prevention of Influenza H7N9 Disease in Adults 50 to 70 Years Old
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: URMC 14-004
Record Dates: First submitted 2014-10-22; First posted 2014-10-24 (Estimated); Last update posted 2017-04-19 (Actual); Status verified 2017-04

CONDITIONS: Influenza A Virus, H7N9 Subtype

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- H7N9 live attenuated vaccine & inactivated subvirion H7N9 vac. (Experimental): Participants will receive one dose of the H7N9 vaccine at Days 0 and 28. They will receive one dose of the inactivated subvirion H7N9 vaccine on Day 98.
  Interventions: Biological: H7N9 Anhui 2013/AA ca; Biological: Inactivated subvirion H7N9 vaccine

INTERVENTIONS:
Biological: H7N9 Anhui 2013/AA ca — 10^7.0 fluorescent focus units (FFU); 0.5 mL of vaccine will be delivered as a nasal spray by an Accuspray device (0.25 mL per nostril)
  Other Names: H7N9 (6-2) AA ca recombinant vaccine; A/Anhui/1/2013 (H7N9) x A/Ann Arbor/6/60 ca; H7N9 A/Anhui/13 ca pLAIV
Biological: Inactivated subvirion H7N9 vaccine — 30 mcg
  Other Names: H7N9 pIIV

SUMMARY:
H7N9 viruses have caused an outbreak of severe respiratory disease in 2013-2014 in China that affected many older adults. This study will evaluate the safety of and immune response to a live attenuated H7N9 vaccine in adults 50 to 70 years old.

DETAILED DESCRIPTION:
H7N9 viruses caused an outbreak of severe respiratory disease in China in 2013-2014, which was associated with severe respiratory illness, acute respiratory distress syndrome (ARDS), intensive care unit (ICU) admissions, and death. The outbreak affected older adults and highlighted the need for a vaccine that is effective in this population. Prior studies have demonstrated the safety and immunogenicity of a vaccination regimen in which administration of the experimental H7N9 vaccine (H7N9 Anhui 2013/AA ca) was followed by an H7N9 inactivated vaccine in younger adults. This study will evaluate the safety and immunogenicity of a similar vaccination regimen in healthy adults, 50 to 70 years old, who are H7N9 seronegative.

Participants will be admitted to the inpatient unit 2 days before they will receive their first vaccination with the H7N9 Anhui 2013/AA ca vaccine. All participants will receive one dose of the H7N9 vaccine, delivered as a nasal spray, on Day 0. While in the inpatient unit, study procedures will include physical examinations, medical history reviews, nasal swabs, and blood and urine collections. On Day 9, participants will be discharged from the inpatient unit provided they meet certain medical criteria. If not, they will remain in the isolation unit until the criteria are met.

On Day 26, participants will be readmitted to the inpatient unit, and on Day 28, they will receive one dose of the H7N9 vaccine delivered as a nasal spray. Participants will remain in the inpatient unit until Day 37 and will take part in all of the same study procedures that occurred during the first inpatient stay. On Day 56, all participants will attend a study visit for a blood collection and nasal swab. On Day 98, all participants will receive one dose of the inactivated subvirion H7N9 vaccine. They will attend study visits on Days 101, 105, 112, 126, 154, and 180, which will include the same study procedures that occurred during the inpatient visits.

ELIGIBILITY:
Inclusion Criteria:

* Adult males and non-pregnant females between 50 years and 70 years of age inclusive. Children will not be recruited or enrolled in this study because they are not in the apparent risk group, and for safety considerations and because of the need for isolation.
* Are in good health, as determined by medical history and targeted physical examination to ensure any existing medical diagnoses or conditions (except those exclusionary) are stable. More information on this criterion can be found in the protocol.
* Agree to storage of blood specimens for future research
* Available for the duration of the trial. Participants must be willing and able to remain within the Isolation Unit for the specified duration of confinement.
* Willingness to participate in the study as evidenced by signing the informed consent document
* Female participants of child-bearing potential must agree to use effective birth control methods for the duration of the study (for example, pharmacologic contraceptives including oral, parenteral, and transcutaneous delivery; condoms with spermicide; diaphragm with spermicide; intrauterine device; abstinence from heterosexual intercourse; surgical sterilization). All female participants will be considered being of child-bearing potential except those who have undergone hysterectomy and those in whom menopause occurred at least 1 year prior to the study.
* Agrees not to participate in another clinical trial with an investigational product for the entire duration of the study

Exclusion Criteria:

* Pregnancy as determined by a positive human choriogonadotropin (beta-HCG) test
* Evidence of clinically significant neurologic, cardiac, pulmonary, hepatic, rheumatologic, autoimmune, or renal disease by history, physical examination, and/or laboratory studies including urine testing. Alanine aminotransferase (ALT) levels greater than 2 times the upper normal limit will be exclusionary at baseline, prior to vaccination.
* Any current illness requiring daily medication other than the following: vitamins, birth control, anti-hypertensive medication, antihistamines, anti-depressant medication, cholesterol lowering medication, treatment for gastroesophageal reflux disease (GERD), and thyroid medication unless approved by the principal investigator.
* Behavioral or cognitive impairment or psychiatric disease that in the opinion of the investigator affects the ability of the participant to understand and cooperate with the study protocol
* Previous enrollment in an H7 or H9 influenza vaccine trial or in any study of an avian influenza vaccine
* Seropositive to the H7N9 influenza A virus (serum HAI titer greater than 1:8)
* Positive urine drug toxicology test indicating narcotic use/dependency
* Have medical, occupational, or family problems as a result of alcohol or illicit drug use during the past 12 months
* Other condition that in the opinion of the investigator would jeopardize the safety or rights of a participant in the trial or would render the participant unable to comply with the protocol
* History of anaphylaxis to any components of the H7N9 vaccines
* Allergy to oseltamivir as determined by participant report
* Current diagnosis of asthma or reactive airway disease (within the past 2 years)
* History of Guillain-Barré Syndrome
* Positive ELISA and confirmatory Western blot tests for human immunodeficiency virus-1 (HIV-1)
* Positive ELISA and confirmatory test (e.g., recombinant immunoblot assay) for hepatitis C virus (HCV)
* Positive hepatitis B virus surface antigen (HBsAg) by ELISA
* Known immunodeficiency syndrome
* Use of corticosteroids (excluding topical preparations) or immunosuppressive drugs within 30 days prior to vaccination
* Receipt of a live vaccine within 4 weeks or a killed vaccine within 2 weeks prior to study vaccination
* History of asplenia
* Receipt of blood or blood-derived products (including immunoglobulin) within 6 months prior to study vaccination
* Current smoker unwilling to stop smoking for the duration of the inpatient stay. A current smoker includes anyone stating they currently smoke or use any amount of a tobacco product, including electronic cigarettes. After admission to the unit, nicotine patches will be provided to current smokers who request them for the inpatient portion of the study.
* Travel to the Southern Hemisphere within 14 days prior to study vaccination
* Travel on a cruise ship within 14 days prior to study vaccination
* Receipt of another investigational vaccine or drug within 30 days prior to study vaccination
* Allergy to eggs, egg products, or formaldehyde

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2014-10; Primary Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Frequency of vaccine-related reactogenicity events (REs) that occur during the acute monitoring (inpatient) phase of the study | Measured through Day 37
Area under the curve (AUC) of nasal virus shedding after each dose of vaccine | Measured through Day 180
  Assessed by liquid titration of nasal secretions on Madin Darby canine kidney (MDCK) cells at 33°C
Development of serum antibody assessed by either hemagglutination inhibition (HAI) or microneutralization (MN) assays following the H7N9 pLAIV or pIIV doses | Measured through Day 180

SECONDARY OUTCOMES:
Development of a significant increase in nasal secretion hemagglutinin (HA)-specific antibody assessed by enzyme-linked immunosorbent assay (ELISA) | Measured through Day 180
Development of greater than 200 influenza-specific interferon-gamma-secreting cells per million lymphocytes as assessed by enzyme-linked immuno spot assay (ELISPOT) on Day 28 after immunization | Measured through Day 28
Detection of influenza-specific IgG or IgA secreting B cells on Day 7 following pLAIV vaccination assessed by antibody secreting cells (ASC) assay | Measured through Day 7

CONTACTS AND LOCATIONS:
Overall Officials: John Treanor, MD, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester Medical Center, Rochester, New York, United States

REFERENCES:
- [Derived] Sobhanie M, Matsuoka Y, Jegaskanda S, Fitzgerald T, Mallory R, Chen Z, Luke C, Treanor J, Subbarao K. Evaluation of the Safety and Immunogenicity of a Candidate Pandemic Live Attenuated Influenza Vaccine (pLAIV) Against Influenza A(H7N9). J Infect Dis. 2016 Mar 15;213(6):922-9. doi: 10.1093/infdis/jiv526. Epub 2015 Dec 9. PMID 26655841